CLINICAL TRIAL: NCT03140670
Title: A Phase 2, Open Label Study of Rucaparib in Patients With Advanced Pancreatic Cancer and a Known Deleterious Germline or Somatic BRCA or PALB2 Mutation
Brief Title: Maintenance Rucaparib in BRCA1, BRCA2 or PALB2 Mutated Pancreatic Cancer That Has Not Progressed on Platinum-based Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 05217
Record Dates: First submitted 2017-05-03; First posted 2017-05-04 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RUCAPARIB

INTERVENTIONS:
Drug: RUCAPARIB — Rucaparib is a PARP inhibitor used as an anti-cancer agent. Rucaparib is a first-in-class pharmaceutical drug targeting the DNA repair enzyme poly-ADP ribose polymerase-1.

SUMMARY:
The main purpose of this study is to look at the effectiveness, safety, and antitumor activity (preventing growth of the tumor) of the experimental study drug rucaparib (also known as CO-338) on subjects and on their pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma with locally advanced or metastatic disease
* ≥18 years of age.
* Eastern Cooperative Oncology (ECOG) performance status of 0 to 1.
* Patients may have previously failed non-platinum containing therapy or may never have previously progressed on treatment.
* Patients must be on treatment with platinum-based (cisplatin, oxaliplatin or carboplatin) treatment for locally advanced or metastatic pancreatic cancer and have received a minimum of 16 weeks of therapy without evidence of disease progression based on the investigator's opinion.
* Discontinuation of the platinum component of the regimen for chemotherapy-related toxicity is permissible provided the patient has previously received at least 16 weeks of platinum-based therapy without evidence of disease progression ≤8 weeks after treatment with the platinum agent
* Documented deleterious BRCA1/2 or PALB2 mutation (germline or somatic) as assessed by CLIA certified laboratory. Variants that are considered to be non-detrimental ("Variants of uncertain significance", "Variants of unknown significance", "Variant, favor polymorphism" or "benign polymorphism" etc) are not sufficient for study entry.
* Measurable disease is not required for enrollment.
* Adequate organ function confirmed by the following laboratory values obtained ≤7 days prior to the first day of rucaparib:

  1. Absolute neutrophil count (ANC) ≥1.5 x 109/L
  2. Platelets>100 x 109/L
  3. Hemoglobin≥9g/dL
  4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN)
  5. Total bilirubin ≤1.5 x ULN; if liver metastases or metabolic disorder such as Gilbert's syndrome, then ≤2.5 x ULN.
  6. Serum creatinine ≤1.5 x ULN or estimated glomerular filtration rate (GFR) ≥45 mL/min using Cockcroft Gault formula.

Exclusion Criteria

* Prior treatment with a PARP inhibitor
* Patients who have demonstrated resistance to platinum agents (e.g. oxaliplatin, cisplatin) are not eligible to participate in this study
* Clinical evidence of uncontrolled malabsorption and/or any other gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with the absorption of rucaparib
* Acute infection requiring intravenous antibiotics, antiviral or antifungal agents during the 14 days prior to first dose of rucaparib
* Symptomatic or untreated CNS metastases.
* Expected life expectancy of <12 weeks as determined by the investigator.
* For fertile patient (female able to become pregnant or male able to father a child), refusal to use effective contraception during the period of the trial and for 6 months after the last dose of rucaparib.
* Received any systemic treatment for pancreatic cancer ≤14 days prior to first dose of rucaparib.
* Non-study related minor surgical procedure ≤5 days, or major surgical procedure ≤21 days, prior to the first dose of rucaparib; in all cases, patients must be sufficiently recovered and stable before treatment administration.
* Active drug or alcohol use or dependence that would interfere with study compliance.
* Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and, in the opinion of the investigator, would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Reiss Binder, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Brown TJ, Yablonovitch A, Till JE, Yen J, Kiedrowski LA, Hood R, O'Hara MH, Teitelbaum U, Karasic TB, Schneider C, Carpenter EL, Nathanson K, Domchek SM, Reiss KA. The Clinical Implications of Reversions in Patients with Advanced Pancreatic Cancer and Pathogenic Variants in BRCA1, BRCA2, or PALB2 after Progression on Rucaparib. Clin Cancer Res. 2023 Dec 15;29(24):5207-5216. doi: 10.1158/1078-0432.CCR-23-1467. PMID 37486343
- [Derived] Reiss KA, Mick R, O'Hara MH, Teitelbaum U, Karasic TB, Schneider C, Cowden S, Southwell T, Romeo J, Izgur N, Hannan ZM, Tondon R, Nathanson K, Vonderheide RH, Wattenberg MM, Beatty G, Domchek SM. Phase II Study of Maintenance Rucaparib in Patients With Platinum-Sensitive Advanced Pancreatic Cancer and a Pathogenic Germline or Somatic Variant in BRCA1, BRCA2, or PALB2. J Clin Oncol. 2021 Aug 1;39(22):2497-2505. doi: 10.1200/JCO.21.00003. Epub 2021 May 10. PMID 33970687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed at the Abramson Cancer Center at the University of Pennsylvania. Patients were enrolled from September 2017 through October 2019.
Pre-assignment Details: Of 46 enrolled patients, 42 patients were evaluable for efficacy analysis. Thus, the enrollment goal was met, per the Protocol.
Groups:
- Single Arm: RUCAPARIB: Rucaparib was used as a maintenance therapy for eligible PDAC patients who received at least 16 weeks of platinum-based chemotherapy without evidence of platinum resistance. Chemotherapy was discontinued and patients received rucaparib 600 mg orally twice a day until progression.
Period: Overall Study
Arm/Group | Single Arm
Started | 46
Completed | 42
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Patients had locally advanced or metastatic pancreatic cancer (neuroendocrine excluded); and had a confirmed pathogenic or likely pathogenic germline or somatic variant in BRCA1, BRCA2, or PALB2. Patients were required to have received at least 16 weeks of platinum-based chemotherapy for locally advanced or metastatic disease without evidence of platinum resistance.
Arm/Group | Single Arm
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] — 18 years of age and older
  years | 61.5 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 40
  Black or African American | 2
  Asian | 0
  Hispanic or Latino | 3
Mutations at baseline: gBRCA2, gBRCA1, gPALB2, sBRCA2. [Count of Participants; unit: Participants]
  Germline BRCA1 | 7
  Germline BRCA2 | 27
  Germline PALB2 | 6
  Somatic BRCA2 | 2
Tumor histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 40
  Acinar | 1
  Squamous cell carcinoma | 1
Disease stage at study start [Count of Participants; unit: Participants]
  Metastatic | 40
  Locally advanced | 2
Platinum treatment duration [Count of Participants; unit: Participants]
  4-6 months | 26
  6-12 months | 5
  More than 12 months | 3
  Less than 4 months | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 6 Months (PFS6)
Description: Time from initiation of rucaparib until progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Only if absolute increase is equal to or greater than 5mm.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 42
Percentage of participants | 59.5 [44.6 to 74.4]

2. Secondary Outcome: Overall Survival
Description: Time from initiation of rucaparib until death or last follow-up
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm
Number analyzed (Participants) | 42
Months | 23.5 [20 to 27]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Confirmed Complete Response or Partial Response according to RECIST v1.1. Complete Response (CR) is defined as tumor burden reduced to 0.0 mm or lymph node lesions are smaller than 10mm. Partial Response (PR), tumor burden decreased by greater than 30% but not CR. Overall Response Rate (ORR) is defined as confirmed CR or PR.
Time Frame: 24 months
Population: Evaluable patients with measurable disease
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 36
Percentage of participants | 41.7 [25.5 to 59.2]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Confirmed complete response, partial response, or stable disease lasting for at least 16 weeks
Time Frame: 24 months
Population: Evaluable patients with measurable disease
Measure: Number (95% Confidence Interval); unit: Percentage of evaluable patients
Arm/Group | Single Arm
Number analyzed (Participants) | 36
Percentage of evaluable patients | 66.7 [49 to 81.4]

5. Secondary Outcome: Duration of Response (DOR)
Description: Time from initial response to progression or death from any cause
Time Frame: 24 months
Population: Evaluable patients with measurable disease
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm
Number analyzed (Participants) | 36
Months | 17.3 [8.8 to 25.8]

6. Secondary Outcome: Toxicity at Least Possibly Related to Rucaparib
Description: Toxicity of rucaparib as maintenance therapy was assessed by examining Adverse Events (AEs) that were at least possibly related to the drug treatment. AEs were classified and graded according to the NCI Common Terminology Criteria of Adverse Events, version 4.1.
Time Frame: 24 months
Measure: Number; unit: Percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 46
Percentage of participants
  Anemia | 74
  Nausea | 48
  Increased ALT | 47
  Fatigue | 45
  Thrombocytopenia | 39
  Dysgeusia | 37

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events (AEs) were classified and graded according to the NCI Common Terminology Criteria of Adverse Events, version 4.1.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 33/42
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=42)
Hepatic dysfunction (Hepatobiliary disorders) | 1 — Included Grade 2 elevated bilirubin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT03140670/Prot_SAP_000.pdf